CLINICAL TRIAL: NCT02936284
Title: Enhancing Alternatives to Eating in Infancy
Brief Title: Infant Environment Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Leonard Epstein, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1134699-1-75860; 1R01HD087082-01A1 (NIH)
Record Dates: First submitted 2016-08-19; First posted 2016-10-18 (Estimated); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Infant Development; Motivation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music Enhancement (Experimental): 37 weekly Music Together classes for one year, then 12 monthly Music Together classes the following year.
  Interventions: Behavioral: Music Enhancement
- Play Date (Active Comparator): 37 weekly group Play Date sessions for one year, then 12 monthly group Play Date sessions the following year.
  Interventions: Behavioral: Play Date

INTERVENTIONS:
Behavioral: Music Enhancement
  Arms: Music Enhancement
Behavioral: Play Date
  Arms: Play Date

SUMMARY:
This study evaluates the effect of a music enhancement program to strengthen the motivation to engage in music related behaviors rather than eating in infants who are high in motivation to eat. Half the participants will participate in a Music Together Program, while the other half will participate in a Play Date control. For both groups, participants will attend 34 weekly sessions for one year, and 12 monthly sessions the next year, in 6 cohorts.

DETAILED DESCRIPTION:
Obesity is a disorder of positive energy balance in which energy intake exceeds energy expenditure. The motivation to eat is a basic human need, which is present at birth. One factor that may lead to increased energy intake is the imbalance between the motivation to eat and the motivation to engage in other behaviors. The motivation to eat versus engaging in other behaviors can be operationalized as the relative reinforcing value of eating versus alternative behaviors.

A strong motivation to eat instead of engaging in alternative behaviors has been related to increased energy intake in adults. The motivation to eat is cross-sectionally and prospectively related to obesity in children, adolescents, and adults, and cross-sectionally related to weight status in infants. Shifting the balance from high motivation to eat to increased motivation to engage in alternative behaviors can reduce energy intake, and may be protective against weight gain.

A structured program to enhance music engagement in infants who are strongly motivated to eat can shift their choice from food to music. This study will expand on this preliminary research and examine long-term effects of this intervention in infants who are highly motivated to eat.

ELIGIBILITY:
Inclusion Criteria:

* High food reinforcement

Exclusion Criteria:

* born preterm (<37 weeks gestation)
* a low birth weight (< 2500 grams)
* known developmental delay(s)
* subject's mother was < 18 years old at the time of pregnancy
* not yet eating finger foods

Ages: 9 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2016-11; Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Epstein, Ph.D, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon request to PI

REFERENCES:
- [Derived] Smith AR, McGregor CM, Carr K, Epstein LH, Serwatka C, Paluch R, Piazza J, Shisler S, Kong KL. The impact of a music enrichment program during infancy and early toddlerhood on effortful control at age 3: A preliminary investigation. Infancy. 2024 Jan-Feb;29(1):72-79. doi: 10.1111/infa.12563. Epub 2023 Oct 12. PMID 37823562
- [Derived] Kong KL, Eiden RD, Morris KS, Paluch RA, Carr KA, Epstein LH. Reducing relative food reinforcement of infants using a music enrichment program: a randomized, controlled trial. Am J Clin Nutr. 2022 Dec 19;116(6):1642-1653. doi: 10.1093/ajcn/nqac209. PMID 36250608
- [Derived] Kong KL, Shisler S, Eiden RD, Anzman-Frasca S, Piazza J. Examining the Relationship between Infant Weight Status and Parent-Infant Interactions within a Food and Nonfood Context. Child Obes. 2022 Sep;18(6):422-432. doi: 10.1089/chi.2021.0126. Epub 2022 Jan 12. PMID 35021890

RESULTS

PARTICIPANT FLOW:
Groups:
- Music Enhancement: 37 weekly Music Together classes for one year, then 12 monthly Music Together classes the following year.
  Music Enhancement
- Play Date: 37 weekly group Play Date sessions for one year, then 12 monthly group Play Date sessions the following year.
  Play Date
Period: Overall Study
Arm/Group | Music Enhancement | Play Date
Started (Participant units are mother-infant dyads, so 47 dyads consisting of 1 mother and 1 child started in each group in the study) | 47 | 47
Completed | 37 | 38
Not Completed | 10 | 9
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 7 | 8

BASELINE CHARACTERISTICS:
Population: Mother-infant dyads
Groups:
- Total: Total of all reporting groups
Arm/Group | Music Enhancement | Play Date | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: months] | 12.1 (1.7) | 11.9 (2.1) | 12.0 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Infant sex
  Participants
    Female | 24 | 23 | 47
    Male | 21 | 22 | 43
Sex: Female, Male [Count of Participants; unit: Participants] — Parent sex
  Participants
    Female | 45 | 45 | 90
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Infant Ethnicity
  Participants
    Hispanic or Latino | 4 | 2 | 6
    Not Hispanic or Latino | 41 | 43 | 84
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Mother Ethnicity
  Participants
    Hispanic or Latino | 3 | 0 | 3
    Not Hispanic or Latino | 42 | 45 | 87
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Infant Race
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 2 | 2
    White | 35 | 37 | 72
    More than one race | 9 | 4 | 13
    Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Mother Race
  Participants
    American Indian or Alaska Native | 0 | 2 | 2
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 2 | 3
    White | 39 | 39 | 78
    More than one race | 4 | 0 | 4
    Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants] — Buffalo, NY. Both members of the dyad were enrolled from the same region
  participants
    United States | 45 | 45 | 90
Weight-for-length z-score [Mean (Standard Deviation); unit: z-score] — Weight for length is a measure of an infant (child under 5-years of age) height (cm) and weight (kg) scored using the World Health Organization (WHO) infant growth chart. Overweight cut-offs at a z-score between 1.0-1.99 and obese cut offs are at a z-score of >=2.0
  z-score | -0.96 (1.63) | -0.55 (1.72) | -0.755 (1.68)
Mother Age [Mean (Standard Deviation); unit: years] | 31.6 (3.9) | 33.2 (4.1) | 32.4 (4.0)
Household income, categorical [Count of Participants; unit: Participants]
  <$50,000/year | 7 | 9 | 16
  >=$50,000/year | 35 | 35 | 70
  No Response | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Infant Food Reinforcing Proportion
Description: Food reinforcing proportion measures responding for food / total responding for both food and music as a proportion score. Scores range from 0 to 1.0 and higher scores indicate more responding for food than for non-food alternative reinforcer of music. Means reported here are estimated from the mixed-model regression analysis
Time Frame: 0-, 3-, 6-, 12-, 24- month
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: proportion food response/total response
Arm/Group | Music Enhancement | Play Date
Number analyzed (Participants) | 45 | 45
proportion food response/total response
  Baseline food reinforcing proportion | 0.66 (0.19) | 0.64 (0.19)
  3-month food reinforcing proportion | 0.53 (0.20) | 0.54 (0.22)
  6-month food reinforcing proportion | 0.48 (0.20) | 0.58 (0.23)
  12-month food reinforcing proportion | 0.44 (0.22) | 0.63 (0.23)
  24-month food reinforcing proportion | 0.47 (0.22) | 0.50 (0.22)
Statistical Analysis 1: Comparison: Music Enhancement vs Play Date; Test type: Superiority; p = 0.016, Mixed Models Analysis; mixed effect regression model including covariates: child sex, child birth weight, breastfeeding duration, percent class attendance and covid grouping; Mean Difference (Net) = 0.196 — difference between music and play group change

2. Secondary Outcome: Infant 24-Hour Dietary Recall- Change in Energy Intake
Description: Energy intake was measured using a 24-recall with the parent and average kcals are reported. One participant was excluded for underreporting
Time Frame: 0-, 12-, 24- month
Population: one participant excluded for underreporting
Measure: Mean (Standard Error); unit: kilocalories
Arm/Group | Music Enhancement | Play Date
Number analyzed (Participants) | 44 | 45
kilocalories
  Baseline child average kcal | 914.2 (33.5) | 898.2 (33.8)
  12-month child average kcal | 1163.5 (46.7) | 1092.2 (52.1)
  24-month child average kcal | 1247.8 (42.9) | 1201.9 (43.9)
Statistical Analysis 1: Comparison: Music Enhancement vs Play Date; mixed effect regression analysis, unstructured covariance, no covariates. Reporting group x time interaction; Test type: Superiority; p = 0.70, Mixed Models Analysis; Mean Difference (Net) = 29.9 — music group vs. play group baseline to 24 months

3. Secondary Outcome: Change in Infant Weight-for-length Z-score
Description: Weight for length is a measure of an infant (child under 5-years of age) height (cm) and weight (kg) scored using the World Health Organization (WHO) infant growth chart. Overweight cut-offs at a z-score between 1.0-1.99 and obese cut offs are at a z-score of >=2.0
Time Frame: 0-, 3-, 6-, 12-, 24- month
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: standardized z-score
Arm/Group | Music Enhancement | Play Date
Number analyzed (Participants) | 45 | 45
standardized z-score
  Baseline child z-weight-for-length | 0.5825 (0.6775) | 0.5646 (0.6977)
  3-month child z-weight-for-length | 0.5566 (0.6929) | 0.5417 (0.7345)
  6-month child z-weight-for-length | 0.6650 (0.7023) | 0.5681 (0.7681)
  12-month child z-weight-for-length | 0.6554 (0.7050) | 0.7444 (0.7896)
  24-month child z-weight-for-length | 0.8271 (0.7366) | 0.7275 (0.7452)
Statistical Analysis 1: Comparison: Music Enhancement vs Play Date; mixed-effect regression analysis with covariates: child sex, birth weight, breastfeeding duration, percent class attendance and covid categories; Test type: Superiority; p = 0.540, Mixed Models Analysis; Mean Difference (Net) = 0.073 — increase in weight for length z-score for music group

ADVERSE EVENTS:
Time Frame: Baseline - two years
Description: Adverse events were collected for the children only.
Arm/Group | Music Enhancement | Play Date
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT02936284/Prot_SAP_000.pdf